CLINICAL TRIAL: NCT04552210
Title: Mannose Binding Lectin Gene Polymorphism Versus Microbial Virulence in the Pathogenesis of Vulvovaginal Candidiasis in Egypt
Brief Title: Mannose Binding Lectin Gene Polymorphism Versus Microbial Virulence in the Pathogenesis of Vulvovaginal Candidiasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Other Study IDs: Mannose
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Detection of MBL2 single nucleotide polymorphisms (SNPs):
  The three SNPs in the promoter regions; rs11003125 (L/H), rs7096206 (Y/X), rs7095891 (P/Q), and one SNP rs1800450 (Gly54Asp) present in codon 54 of MBL2 were genotyped using ARMS-PCR (amplification refractory mutation system- PCR)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood sample — Whole blood was collected on EDTA (1mg/ml) to prevent clotting and DNA degradation.

SUMMARY:
The vaginal mucosa is inhabited by both fungal and bacterial microorganisms which normally co-exist with the host in a tightly regulated and commensal manner.

DETAILED DESCRIPTION:
Nevertheless, under certain circumstances, this co-existence can turn into a pathologic state followed by symptomatic disease

ELIGIBILITY:
Inclusion Criteria:

* 1. Married females in the reproductive age period. 2. Females complaining of vaginal discharge (whitish and scanty), itching, dyspareunia, pruritis, and signs of vulvovaginitis ie. erythema.

Exclusion Criteria:

* females who attended the same clinic in the same period, matched the cases regarding the age group, without having Candida infection as confirmed by culture of vaginal swabs.

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female with candidal infection
Study Population: Married females in the reproductive age period. 2. Females complaining of vaginal discharge (whitish and scanty), itching, dyspareunia, pruritis, and signs of vulvovaginitis ie. erythema.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
the number of women who have mutation in MBL2 gene polymorphism | a month
  women who have mutation in MBL2 gene polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah, Giza, Egypt